CLINICAL TRIAL: NCT00519454
Title: Estrogen and Gender Biased Autoimmunity in Systemic Lupus Erythematosus
Brief Title: Estrogen and Gender Biased Autoimmunity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Center for Rheumatic Disease, Allergy, & Immunology (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Nabih I Abdou, Center for Rheumatic Disease Allergy & Immunology
Other Study IDs: 05-024
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Estrogen receptors; T cells; Hormones; Female adult SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Female Lupus patients: Females who are still childbearing age, not on hormones, with Systemic Lupus Erythematosus, still cycling.
  Interventions: Other: Peripheral lab draws

INTERVENTIONS:
Other: Peripheral lab draws — 100ml blood for analysis, taken no more than 4 times in one year.

SUMMARY:
This study involves research to investigate how estrogen affects women of childbearing age and its correlation to Systemic Lupus Erythematosus. The findings from this study might help determine how body cells, called T Cells, react to estrogen. The study will seek to determine if cells from women with Lupus, react differently from cells in persons without Lupus. We will attempt to identify genetic factors that determine the effects of estrogen on Lupus cells.

DETAILED DESCRIPTION:
This is a 3-year study. The total number of subjects enrolled will depend on the results obtained. The subjects will be at least 18 years of age and pre-menopausal. Exclusion to include pregnant women, and all subjects are told not to get pregnant while on study. Also, they cannot take hormones by mouth or patch while on study. The study can include healthy subjects as well. Blood will be drawn (120 ml) four times a year, randomly.

ELIGIBILITY:
Inclusion Criteria:

* female subjects with Lupus, and female subjects without Lupus. age at least 18, not pregnant and not planning to get pregnant.

Exclusion Criteria:

* Pregnant or planning to get pregnant. On hormone replacement, or birth control of any kind.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female subjects with SLE and still cycling, not on hormones, compared to normal controls, female subjects still cycling, also not on hormones and not diagnosed with SLE.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2005-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nabih I Abdou, MD, PhD, Principal Investigator — The Center for Rheumatic Disease, Allergy and Immunology
Locations (1):
- The Center for Rheumatic Disease, Allergy and Immunology, Kansas City, Missouri, United States